CLINICAL TRIAL: NCT02068950
Title: Feasibility of a 12-week Progressive Resistance Training Program in Head and Neck Cancer Patients During Concurrent Radiochemotherapy - a Pilot Trial
Brief Title: Progressive Resistance Training Program in Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Julie Gehl, Senior Consultant, ph.d., Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HH1401
Record Dates: First submitted 2014-02-13; First posted 2014-02-21 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer; Concurrent chemoradiotherapy; Progressive resistance training; Exercise; Feasibility; Weight loss; LBM; Body composition
MeSH Terms: conditions — Head and Neck Neoplasms; Motor Activity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Progressive resistance training (Other): 12 weeks, 3 sessions per week, 7 exercises (leg press, leg curl, hamstring curl, chest press, lateral pull down, sit-ups and back extensions). In general 2-3 sets of 8-15 repetitions will be performed following a progression plan starting with more repetitions at lower intensity progressing to fewer repetitions at higher intensity during the 12-week period (American College of Sports Medicine Position Stand).
  Interventions: Behavioral: Progressive resistance training

INTERVENTIONS:
Behavioral: Progressive resistance training — A 12-week, supervised, group based, progressive resistance training program involving the major muscle groups of the body will be tested. Details of the program: 12 weeks, 3 sessions per week, 7 exercises (leg press, leg curl, hamstring curl, chest press, lateral pull down, sit-ups and back extensions). In general 2-3 sets of 8-15 repetitions will be performed following a progression plan starting with more repetitions at lower intensity progressing to fewer repetitions at higher intensity during the 12-week period (American College of Sports Medicine Position Stand)

SUMMARY:
The purpose of this study is to evaluate the feasibility of a 12-week progressive resistance training (PRT) during concurrent chemoradiotherapy in head and neck cancer patients compared to usual care.

DETAILED DESCRIPTION:
12 patients with head and neck cancer will be recruited to this trial. Entering a 12-week PRT program which will start one week before radiotherapy. The tested training program is a 12-week, supervised, group based, progressive resistance training program involving the major muscle groups of the body. The program has previously been found to successfully restore the loss of lean body mass (LBM) in head and neck cancer patients post-treatment. A group based approach will be used to facilitate a social and motivating training environment for the patients. This approach has previously been used for exercise interventions for lung cancer patients at our facility, and was highly appreciated by the patients.

In addition to baseline data (height, tumor stage, performance status, etc), the following parameters will be registered on a weekly basis: Weight, patient reported side effects, as well as a questionnaire on amount of physical activity and food intake.

Physical function and strength will be tested at baseline, after the course of chemoradiotherapy and at the end of the 12-week PRT programme, and at 2, 5, 9 and 13 months follow-up. At similar time points dual energy x-ray absorptiometry (DXA) scans for body composition will be performed using a Lunar iDXA (GE Healthcare).

Blood samples will be drawn at baseline, an additional three times during the first 6 weeks and then weekly in relation to training sessions, and at 2, 5, 9 and 13 months follow-up.

Patient reported quality of life (EORTC Quality of Life Questionaire (QLQ)-C30 and QLQ-H&N35) will be registered at baseline, after 12-weeks PRT and during 5 and 13 months follow-up.

Study duration is expected to be 7 months for the pilot-trial, with a follow-up of additional 13 months after the last patient has completed the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck squamous cell carcinoma
* Candidates for concomitant chemoradiotherapy according to Danish Head and Neck Cancer Group (DAHANCA) guidelines.
* Performance status 0-1
* Expected to be able to complete the intervention, i.e. no major comorbidities or social issues that could compromise attendance.
* At least 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Feasibility | up to 7 months
  The feasibility outcomes will be inclusion rate defined as the number of patients recruited from the number of eligible patients and completion rate defined as the number of participants able to complete the intervention.
  Adherence to the exercise intervention will be evaluated via patient-reported training logs.

SECONDARY OUTCOMES:
Change in LBM | up to 20 months
  Whole body LBM will be determined using dual energy x-ray absorptiometry (DXA).
Weight loss | up to 20 months
  Patient will be weighed weekly during the 12-week PRT program; afterwards at each follow-up (2, 5, 9, and 13 months)
Number of patients with side-effects to treatment | up to 7 months
  Side-effects will be registered using Common Terminology Criteria for Advers Events v4.0 (CTCAE).
Quality of Life | Up to 20 months
Change in physical function and strength | Up to 20 months
  Change in muscle strength will be evaluated by 1 repetition maximum test (1RM) measured in kg.
  Change in muscle power will be evaluated by Nottingham Power Rig and measured in watts and watt/kg.
  Change in physical function will be evaluated by 30 second sit-to-stand test, arm curl test and stair climbing.

OTHER OUTCOMES:
Muscle biopsies | up to 7 months
  In order to establish energy-reserves in the muscles
Blood samples | Up to 20 months
  In order to identify systemic factors released during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, ph.d., Principal Investigator — Herlev Hospital
Locations (1):
- Dept. of Oncology, Herlev, Denmark